CLINICAL TRIAL: NCT01072656
Title: Deep Brain Stimulation for Thalamic Pain Syndrome
Brief Title: Safety Study of Deep Brain Stimulation to Manage Thalamic Pain Syndrome
Acronym: DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andre Machado (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Andre Machado, Staff Physician, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AGM-001; 1DP2OD006469-01 (NIH)
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Active Comparator): Active stimulation and programmed to the settings found to be optimal during the titration process.
  Interventions: Device: Deep Brain Stimulation for Thalamic Pain Syndrome
- Control group (Sham Comparator): IPG is set to ON but the voltage is set to 0V.
  Interventions: Device: Deep Brain Stimulation for Thalamic Pain Syndrome

INTERVENTIONS:
Device: Deep Brain Stimulation for Thalamic Pain Syndrome — Patients will be randomized in a 1:1 ratio to one of two groups: the Treatment Group (active stimulation and programmed to the settings found to be optimal during the titration phase) and the Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V). In order to prevent too many patients from being randomized to ON or to sham early in the study, we will use, for the first 4 patients, randomization blocks of four or six. In this fashion, the first four consecutive patients will have two patients randomized to the Treatment Group and two patients in the Control Group. In the same fashion, the final six patients will have three patients randomized to the treatment group and three patients to the control group.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Deep Brian Stimulation (DBS) of the ventral capsular/ventral striatal as a treatment for patients with Thalamic Pain Syndrome (TPS). The central hypothesis to be tested in this investigation is that VC/VS stimulation will modulate the affective component of TPS and, consequently, improve pain related disability.

DETAILED DESCRIPTION:
This is a pilot clinical study of the therapeutic benefits of ventral capsular/ventral striatal deep brain stimulation (DBS) as a treatment for 10 patients with medically refractory thalamic pain syndrome. Patients to be enrolled under this protocol will have experienced severe pain for more than six months and will be considered medically refractory. Study subjects may have undergone and failed other surgical procedures or interventional procedures. Study subjects will have chronic, medically refractory pain of disabling severity, refractory to treatment attempts with conventional medications. Patients that are enrolled in the study will have bilateral DBS surgery, with implantation of one Medtronic 3391 DBS lead on either side of the brain. These leads will then be connected at first to a single Medtronic PC pulse generator to be implanted in the infraclavicular region on one side. Once the PC pulse generator is depleted, and the patient has completed the blinded phase of the study, the PC pulse generator will be replaced for an RC pulse generator. The RC pulse generator has a battery life of 9 years and is a good option for the open label phase and for continued stimulation after the study is completed. However, the RC is not ideal for the blinded phase because patients may be able to tell if they are receiving active or sham stimulation. For this reason, patients enrolled in this study will receive, initially, the implant with the PC generator. Patients will have at least 6 months of stable chronic pain associated with TPS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of thalamic pain syndrome
* with allodynia or dysesthesia
* with pinprick anesthesia or hypoesthesia on the affected hemibody (anesthesia dolorosa).
* Six months or more of medically refractory severe pain (see below).
* Pain disability reported by the pain index >30 points at the time of enrollment.
* Average daily pain for the past 30 days reported as >5 on a 0-10 scale
* Failure to respond adequately to at least one antidepressant, one anti-seizure medication and one oral narcotic.
* MRI done within one year of the first visit showing a lesion that involves the posterior thalamic region or a lesion in the dorsal or ventral vicinity of the thalamus (i.e. semi oval white matter or brain stem). The lesion will be contralateral to the hemibody affected by chronic pain or will involve cortical-subcortical areas in topography consistent with sensory thalamocortical connections. This will include patients with infarcts in the territory of the middle cerebral artery. A more recent MRI may be required if the patient's condition changed within the previous year.
* Capable of understanding and providing informed consent
* Age ≥ 21 years
* Women of childbearing age must be on regular use of an accepted contraceptive method(s).
* Previous surgical procedures: Patients with severe and refractory thalamic pain syndrome may have undergone other interventional or surgical procedures, as an attempt to alleviate the thalamic pain syndrome. Surgical procedure may include blocks, spinal cord stimulation, thalamic DBS, posterior limb of the internal capsule DBS or periaqueductal gray / periventricular gray DBS, cortical stimulation, peripheral ablative procedures or cerebral ablative procedures. In this study, patients with previously implanted cortical stimulation systems, or spinal and peripheral nervous system stimulation systems may be included. However, patients with previous motor cortex stimulation must have had the cortical stimulation system before being considered a candidate for this protocol. Removal of the cortical stimulation system will not be covered under this protocol. Patients with spinal or peripheral neuromodulation system may be included in the research provided that the implanted systems are compatible with the all research protocols (including fMRI) to be performed during the research. Patients with pervious DBS implants will not be considered candidates.

Exclusion Criteria:

* Not capable of understanding or providing informed consent.
* Aphasia severe enough to limit the consent process or communication between the investigators and the patient. Patients with mild or recovering aphasia may be considered candidates at the discretion of the PI.
* Coagulopathy. Patients will be excluded unless assessed and cleared by hematology
* Inability to stop Coumadin or platelet anti-aggregation therapy for surgery and after surgery. Patients taking these medications will need to discuss the need/risk of continuing these medications with their physicians and the PI or study personnel may contact the treating physician(s) as well to discuss the risks of anticoagulation / antiaggregation therapy discontinuation.
* Uncontrolled hypertension.
* Malignancy with < 5 years life expectancy.
* Major medical co-morbidities: end stage renal failure, heart failure, severe congestive heart disease, severe respiratory problems, liver failure or other significant medical co morbidities.
* Major neurological disorder other than the one that led to the TPS.
* MRI (done within one year of the first visit) with abnormalities other than those associated with the neurological disorder causing TPS.
* Age < 21 years.
* Pregnancy or lack of regular use of contraceptives. Patients who become pregnant after enrollment may be excluded from the study. Patients who become pregnant prior to the surgical implantation of the DBS systems will be excluded from the study.
* Previous ablative intracranial surgery for the management of the TPS.
* Previously implanted with deep brain stimulation system.
* Concurrent enrolment in any other trial / study for TPS.
* Implantable hardware not compatible with MRI or with the study.
* Patients may be excluded from enrollment due to a condition that, in the judgment of the PI, significantly increases risk or reduces significantly the likelihood of benefit from VC/VS DBS.
* Untreated / uncontrolled (severe at the time of enrolment) depression or other psychiatric disorder.
* Bipolar disorder, current PTSD, severe personality disorder, active psychosis, Severe OCD.
* Psychological co-morbidities that indicates higher risk to the patient and / or higher risk of failure.
* Suicide attempt </= 12 months
* Communication of a plan for suicide, prior to implant, should the study treatment fail
* Imminent suicide risk

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2014-08 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre G Machado, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Gopalakrishnan R, Burgess RC, Lempka SF, Gale JT, Floden DP, Machado AG. Pain anticipatory phenomena in patients with central poststroke pain: a magnetoencephalography study. J Neurophysiol. 2016 Sep 1;116(3):1387-95. doi: 10.1152/jn.00215.2016. Epub 2016 Jun 29. PMID 27358316
- [Background] Gopalakrishnan R, Burgess RC, Plow EB, Floden DP, Machado AG. Early event related fields during visually evoked pain anticipation. Clin Neurophysiol. 2016 Mar;127(3):1855-63. doi: 10.1016/j.clinph.2015.11.019. Epub 2015 Dec 5. PMID 26733321
- [Derived] Plow EB, Malone DA Jr, Machado A. Deep brain stimulation of the ventral striatum/anterior limb of the internal capsule in thalamic pain syndrome: study protocol for a pilot randomized controlled trial. Trials. 2013 Jul 31;14:241. doi: 10.1186/1745-6215-14-241. PMID 23902631

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants signed informed consent, 10 participants had surgery, 1 participant dropped the study prior to randomization phase, 9 participants were analyzed.
Groups:
- Active First: active stimulation programmed to the settings found to be optimal during the titration phase
- Sham First: sham stimulation - IPG ON, at 0 Volt
Period: First Intervention
Arm/Group | Active First | Sham First
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Active First | Sham First
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active First | Sham First | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (5.9) | 54 (5.3) | 52 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 50% Improvement in Pain Related Disability (as Assessed by the Pain Disability Index)
Description: Pain Disability Index (PDI) directly measures disability related to the main components of daily life function and has been validated for thalamic pain syndrome. Range is 0 (no disability) to 10 (worst disability). The components are Family/Home Responsibilities, Recreation, Social Activity, Sexual Behavior, Life-support Activity, Occupation, & Self-care. This is an average score of the 3 month period for each Active and Sham phase.
Time Frame: Blinded stimulation phase (3 Months)
Measure: Number; unit: participants
Groups:
- Active Stimulation: Active stimulation and programmed to the settings found to be optimal during the titration process.
  Deep Brain Stimulation for Thalamic Pain Syndrome: Patients will be randomized in a 1:1 ratio to one of two groups: the Treatment Group (active stimulation and programmed to the settings found to be optimal during the titration phase) and the Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V). In order to prevent too many patients from being randomized to ON or to sham early in the study, we will use, for the first 4 patients, randomization blocks of four or six. In this fashion, the first four consecutive patients will have two patients randomized to the Treatment Group and two patients in the Control Group. In the same fashion, the final six patients will have three patients randomized to the treatment group and three patients to the control group.
- Sham Stimulation: IPG is set to ON but the voltage is set to 0V.
  Deep Brain Stimulation for Thalamic Pain Syndrome: Patients will be randomized in a 1:1 ratio to one of two groups: the Treatment Group (active stimulation and programmed to the settings found to be optimal during the titration phase) and the Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V). In order to prevent too many patients from being randomized to ON or to sham early in the study, we will use, for the first 4 patients, randomization blocks of four or six. In this fashion, the first four consecutive patients will have two patients randomized to the Treatment Group and two patients in the Control Group. In the same fashion, the final six patients will have three patients randomized to the treatment group and three patients to the control group.
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 9 | 9
participants | 2 | 0

2. Secondary Outcome: Number of Participants Who Had 50% Improvement in PDI
Description: A 50% improvement in pain related disability (as assessed by the pain disability index) at the end of the open label phase compared to the pre-implantation baseline. The PDI ranges from 0-10 with 0 equaling no disability and 10 equaling worst disability.
Time Frame: 24 months post randomization follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation
Number analyzed (Participants) | 9
Participants | 1

3. Secondary Outcome: Number of Participants Who Would Undergo the Procedure Again.
Description: A positive answer from patients receiving active stimulation at the end of the open label phase of the study to the question: 'would you undergo this procedure again if you were to get the same benefits you experienced?'
Time Frame: End of Open Label Phase (24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation
Number analyzed (Participants) | 9
Participants | 6

4. Secondary Outcome: Number of Patient Who Had >50% Reduction in VAS.
Description: Patients report reduction in the VAS (Visual Analogue Scale Ranging from 0-10, 0 meaning no pain and 10 meaning worst pain imaginable) at the end of the open label phase (24 months post randomization f/u) compared to the pre-implantation baseline.
Time Frame: Baseline and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Stimulation
Number analyzed (Participants) | 9
Participants | 2

ADVERSE EVENTS:
Groups:
- Active Stimulation (Phase V): Active stimulation and programmed to the settings found to be optimal during the titration process.
  Deep Brain Stimulation for Thalamic Pain Syndrome: Patients will be randomized in a 1:1 ratio to one of two groups: the Treatment Group (active stimulation and programmed to the settings found to be optimal during the titration phase) and the Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V). In order to prevent too many patients from being randomized to ON or to sham early in the study, we will use, for the first 4 patients, randomization blocks of four or six. In this fashion, the first four consecutive patients will have two patients randomized to the Treatment Group and two patients in the Control Group. In the same fashion, the final six patients will have three patients randomized to the treatment group and three patients to the control group.
- Sham Stimulation (Phase V): IPG is set to ON but the voltage is set to 0V.
  Deep Brain Stimulation for Thalamic Pain Syndrome: Patients will be randomized in a 1:1 ratio to one of two groups: the Treatment Group (active stimulation and programmed to the settings found to be optimal during the titration phase) and the Control Group (sham stimulation - IPG is set to ON but the voltage is set to 0V). In order to prevent too many patients from being randomized to ON or to sham early in the study, we will use, for the first 4 patients, randomization blocks of four or six. In this fashion, the first four consecutive patients will have two patients randomized to the Treatment Group and two patients in the Control Group. In the same fashion, the final six patients will have three patients randomized to the treatment group and three patients to the control group.
- Phase I-IV: Phase I-IV is time frame of patient consent through surgery just prior to beginning Active v Sham Stimulation Phase.
Arm/Group | Active Stimulation (Phase V) | Sham Stimulation (Phase V) | Phase I-IV
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (Phase V) (N=9) | Sham Stimulation (Phase V) (N=9) | Phase I-IV (N=9)
FOCAL PARTIAL SEIZURE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Complex Partial Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Right Burr Hole Dehiscence (Infections and infestations) | 1 | 0 | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Gastric Ulcer w/out Hemorrhage or Perferation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Post Hemorrhagic Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Kidney Stone Bacteremia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abscessed Tooth (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis from C Diff (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendectomy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (Phase V) (N=9) | Sham Stimulation (Phase V) (N=9) | Phase I-IV (N=9)
Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Patient Fall (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Redness from pulling at scab behind ear at head frame site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hypomania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acid Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (3)
Auditory Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Scalp Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Increased Libido (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Reoccurrence of chronic sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Symptoms from L5-S1 degerative disc disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract complicatoin (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0)
Increased sleep (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increased sensitivity at bottom of feet (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Balance difficulty (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Left ankle pain/giving out (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Itchy scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Attention deficit disorder exacerbation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes III-controlled (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Feels like extremities are in vice (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Outdoor temperature increases pain (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Root canal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Right hand pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening intensity of suicide ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Worsening pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Difficulties concentrating (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Torso extreme tightness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
When left side laying only, torso sweats (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Walking is more ataxic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased pain with DBS turned off (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ED for BP spike (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Edema in right foot (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Carpel tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent leg twitch (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Infection from animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carotid trickling (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes